CLINICAL TRIAL: NCT03677479
Title: Evaluation of Post-extraction Socket Preservation With Camelline Versus Bovine Deproteinized Xenograft (Pilot Trial)
Brief Title: Evaluation of Post-extraction Socket Preservation With Camelline Versus Bovine Deproteinized Xenograft
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ghada Adayil, Teaching Assisstant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: PER123
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Socket Preservation
Keywords: bone grafts; xenograft

STUDY DESIGN:
Intervention Model Description: pilot randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: single blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- socket preservation with camelline bone (Experimental): natural hydroxyapatite derived from camels prepared by investigator
  Interventions: Procedure: socket preservation procedure
- socket preservation with bovine bone (Active Comparator): natural hydroxyapatite derived from cows (Bio-Oss)
  Interventions: Procedure: socket preservation procedure

INTERVENTIONS:
Procedure: socket preservation procedure — socket preservation of post extraction site using bone xenografts
  Other Names: alveolar ridge preservation

SUMMARY:
Alveolar ridge preservation following tooth extraction has the ability to maintain the ridge dimensions and allow the implant placement in an ideal position fulfilling both functional and aesthetic results. Postextraction socket healing commonly results in resorption of the alveolar ridge.

To prevent this clinical situation, different authors have described several surgical procedures, ranging from regenerative techniques for socket preservation to immediate implant placement. Regenerative techniques have been widely tested in controlled and uncontrolled studies with various materials and clinical approaches: bone grafting alone, including autografts, allografts, xenografts, and alloplasts; membrane alone, whether absorbable or not; and membrane in conjunction with grafting.

DETAILED DESCRIPTION:
Various classic studies in the 1960s showed that the resorption process of the postextraction alveolus in both jaws was significantly more pronounced on the buccal aspect. This comes as no surprise, as the buccal surface of the anterior alveolar ridge is commonly thin and fragile. The maxilla tends to exhibit greater reductions in width than in height. The loss of tissue contour takes place mostly during the first 1 to 3 months following tooth extraction. Because the healing patterns of human sockets are unpredictable architecture), then such common procedures as extractions may lead to intraoral situations in which the remaining healed ridge does not allow for an esthetic and functional solution without the aid of significant bone grafting.

ELIGIBILITY:
Inclusion Criteria:

* Teeth with: root fractures, endodontic treatment failures, advanced caries lesions or any other cause that make tooth non-restorable and indicated for extraction.
* Healthy non-smoker patients

Exclusion Criteria:

* Medically compromised patients.
* Pregnant females.
* History of malignancy or radiotherapy/chemotherapy for malignancy in the past 5 years.
* History of active bone metabolic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — patient eligable for implant placement after socket preservation more than 18 years
Enrollment: 10 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
patient-reported outcome | within first week postoperatively
  assessment of post-operative complication( pain, swelling, bleeding, infection)

SECONDARY OUTCOMES:
ridge contour changes | 3 month, 6 month
  dimentional changes after extraction and socket preservation

CONTACTS AND LOCATIONS:
Overall Officials: Manal Hosny, PhD, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided
check with university guidelines for raw data sharing

REFERENCES:
- [Result] Chang PC, Chang HC, Lin TC, Tai WC. Preclinical alveolar ridge preservation using small-sized particles of bone replacement graft in combination with a gelatin cryogel scaffold. J Periodontol. 2018 Oct;89(10):1221-1229. doi: 10.1002/JPER.17-0629. Epub 2018 Aug 29. PMID 30039627